CLINICAL TRIAL: NCT00777387
Title: Cryopreservation of Oocytes: A Randomized Controlled Trial Comparing Slow-freezing to Vitrification
Brief Title: Randomized Controlled Trial Comparing Slow-freezing to Vitrification of Oocytes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Studies emerged that demonstrated the superiority of vitrification
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Principal Investigator, Ellen Greenblatt, Associate Professor, U of T, Samuel Lunenfeld Research Institute, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: oocyte cryopreservation
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Infertility
Keywords: human oocyte cryopreservation; slow-freeze; vitrification
MeSH Terms: conditions — Infertility | interventions — Vitrification

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): slow-freeze
  Interventions: Procedure: slow-freeze
- 2 (Active Comparator): vitrification
  Interventions: Procedure: vitrification

INTERVENTIONS:
Procedure: slow-freeze — Slow-freeze-rapid-thaw procedure of oocytes is characterized by prolonged exposure of the cell to cryoprotectants in a low metabolic state at very low temperatures
  Arms: 1
Procedure: vitrification — Vitrification is the process by which water is prevented from forming ice due to the viscosity of a highly concentrated cryoprotectant cooled at an extremely rapid rate
  Arms: 2

SUMMARY:
Preservation of fertility is limited. Current methods include embryo cryopreservation and while still experimental, ovarian cryopreservation. In single women who are at risk for infertility secondary to cancer or couples who have ethical reasons to avoid embryo cryopreservation, oocyte cryopreservation is an alternative Purpose of study is to compare slow freeze to vitrification of human oocytes. Successful cryopreservation and subsequent thawing programs are characterized by avoiding ice crystal formation.Vitrification, newer alternative to slow freeze method, process by which water is prevented from forming ice.

Our hypothesis is that higher survival rate per oocyte is to be expected in the vitrification group.

DETAILED DESCRIPTION:
Although several reviews of smaller studies of cryoprotectant methodology exist randomized controlled trials,comparing slow-freeze-rapid-thaw procedure to vitrification of oocytes, are not available. The purpose of this study is to compare these two methods of oocyte cryopreservation in human oocytes.

ELIGIBILITY:
Inclusion Criteria:

* 14 or more oocytes at ovum pick up
* age < 38
* bmi < 30

Exclusion Criteria:

-

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2008-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
post-thaw oocyte survival rate | 2 years

SECONDARY OUTCOMES:
fertilization rate | 2 years
cleavage | 2 years
embryo development | 2 years
implantation rate | 2 years
ongoing pregnancy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ellen M Greenblatt, MD, FRCS(C), Study Director — Mount Sinai Hospital, Canada
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Gook DA, Edgar DH. Human oocyte cryopreservation. Hum Reprod Update. 2007 Nov-Dec;13(6):591-605. doi: 10.1093/humupd/dmm028. Epub 2007 Sep 10. PMID 17846105
- [Background] Porcu E, Venturoli S. Progress with oocyte cryopreservation. Curr Opin Obstet Gynecol. 2006 Jun;18(3):273-9. doi: 10.1097/01.gco.0000193015.96275.2d. PMID 16735826
- [Background] Oktay K, Cil AP, Bang H. Efficiency of oocyte cryopreservation: a meta-analysis. Fertil Steril. 2006 Jul;86(1):70-80. doi: 10.1016/j.fertnstert.2006.03.017. PMID 16818031
- [Background] Jain JK, Paulson RJ. Oocyte cryopreservation. Fertil Steril. 2006 Oct;86(4 Suppl):1037-46. doi: 10.1016/j.fertnstert.2006.07.1478. PMID 17008147
- [Background] Byrne J, Fears TR, Gail MH, Pee D, Connelly RR, Austin DF, Holmes GF, Holmes FF, Latourette HB, Meigs JW, et al. Early menopause in long-term survivors of cancer during adolescence. Am J Obstet Gynecol. 1992 Mar;166(3):788-93. doi: 10.1016/0002-9378(92)91335-8. PMID 1550144
- [Background] Falcone T, Attaran M, Bedaiwy MA, Goldberg JM. Ovarian function preservation in the cancer patient. Fertil Steril. 2004 Feb;81(2):243-57. doi: 10.1016/j.fertnstert.2003.06.031. PMID 14967351
- [Background] Porcu E, Fabbri R, Damiano G, Giunchi S, Fratto R, Ciotti PM, Venturoli S, Flamigni C. Clinical experience and applications of oocyte cryopreservation. Mol Cell Endocrinol. 2000 Nov 27;169(1-2):33-7. doi: 10.1016/s0303-7207(00)00348-8. PMID 11155951
- [Background] Sonmezer M, Oktay K. Fertility preservation in young women undergoing breast cancer therapy. Oncologist. 2006 May;11(5):422-34. doi: 10.1634/theoncologist.11-5-422. PMID 16720842
- [Background] Yoon TK, Kim TJ, Park SE, Hong SW, Ko JJ, Chung HM, Cha KY. Live births after vitrification of oocytes in a stimulated in vitro fertilization-embryo transfer program. Fertil Steril. 2003 Jun;79(6):1323-6. doi: 10.1016/s0015-0282(03)00258-9. PMID 12798878